CLINICAL TRIAL: NCT02928263
Title: A Healthcare Cost and Resource Utilization Analysis of Intravenous and Oral Agents in the Treatment of Metastatic Renal Cell Carcinoma
Brief Title: Healthcare Cost and Resource Utilization Related to Metastatic Renal Cell Carcinoma Treatment With Intravenous and Oral Agents
Status: Withdrawn | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-780
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients treated with IV agents: Metastatic renal cell carcinoma patients treated with IV agents
  Interventions: Other: Non-Interventional
- Patients treated with oral agents: Metastatic renal cell carcinoma patients treated with oral agents
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Other

SUMMARY:
A retrospective study to evaluate healthcare cost and resource utilization for patients with metastatic renal cell carcinoma who have been treated with IV or oral agents

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with metastatic renal cell carcinoma
* Prescription/administration of one of the IV or oral agents examined in the study

Exclusion Criteria:

* Patients with other primary cancer diagnosis before RCC diagnosis
* Patients with pregnancy or HIV/AIDS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metastatic RCC patients in the US identified from administrative claim databases
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-05-31 (Estimated); Study Completion 2017-05-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of Healthcare costs for patients treated with oral drugs used in the first-line treatment of Metastatic renal cell carcinoma (mRCC) | Up to 63 months
  All-cause healthcare costs will be calculated in the first-line oral cohort as per-patient-per-month (PPPM) costs.
Composite of Resource Utilization for patients treated with oral drugs used in the first-line treatment of mRCC | Up to 63 months
  Total numbers and rates of inpatient, outpatient, and emergency room visits per patient will be calculated.
Distribution of Healthcare costs for patients treated with IV drugs used in the first-line treatment of mRCC | Up to 63 months
  All-cause healthcare costs will be calculated in the first-line IV cohort as per-patient-per-month (PPPM) costs.
Composite of Resource Utilization for patients treated with IV drugs used in the first-line treatment of mRCC | Up to 63 months
  Total numbers and rates of inpatient, outpatient, and emergency room visits per patient will be calculated.

SECONDARY OUTCOMES:
Medication Possession Ratio (MPR) for patients treated with oral drugs used in the first-line treatment of mRCC | Up to 63 months
  MPR will be calculated for each index drug as the ratio of the sum of the total number of days' supply to the total number of days in the follow-up period.
Medication Possession Ratio (MPR) for patients treated with IV drugs used in the first-line treatment of mRCC | Up to 63 months
  MPR will be calculated for each index drug as the ratio of the sum of the total number of days' supply to the total number of days in the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb, Princeton, New Jersey, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx